CLINICAL TRIAL: NCT00642668
Title: Subcutaneous Treatment of Anemia in Patients With a GFR Below 45 ml/Min/1.73m2 Through Injections With Mircera as Low Frequent as Once Monthly (STABILO)
Brief Title: A Study of Subcutaneous Mircera for the Maintenance Treatment of Participants With Chronic Renal Anemia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML21348
Record Dates: First submitted 2008-03-19; First posted 2008-03-25 (Estimated); Results first posted 2016-07-22 (Estimated); Last update posted 2017-07-05 (Actual); Status verified 2017-05

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — continuous erythropoietin receptor activator

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Methoxy Polyethylene Glycol-Epoetin Beta (Experimental): Participants received methoxy polyethylene glycol-epoetin beta treatment monthly for 36 weeks with an efficacy evaluation period (EEP) during weeks 29-36 and followed by a 4 week follow-up period.
  Interventions: Drug: methoxy polyethylene glycol-epoetin beta

INTERVENTIONS:
Drug: methoxy polyethylene glycol-epoetin beta — 1.2 mcg/kg administered subcutaneously (sc) monthly for 36 weeks (initial recommended dose)
  Other Names: Mircera

SUMMARY:
This single arm study assessed the efficacy and safety of subcutaneous methoxy polyethylene glycol-epoetin beta (Mircera), a continuous erythropoietin receptor activator (C.E.R.A.), for correction and/or maintenance of hemoglobin levels in participants with chronic kidney disease and renal anemia, who were not treated with erythropoiesis-stimulating agents (ESA) or on dialysis. Eligible participants received monthly subcutaneous injections of methoxy polyethylene glycol-epoetin beta at an initial recommended dose of 1.2 micrograms/kilogram (mcg/kg). The anticipated time on study treatment was 3-10 months, and the target sample size was 200 individuals.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants, >=18 years of age;
* Chronic renal anemia;
* No ESA therapy during previous 3 months.

Exclusion Criteria:

* Transfusion of red blood cells during previous 2 months;
* Poorly controlled hypertension requiring hospitalization in previous 6 months;
* Significant acute or chronic bleeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2008-06-30 (Actual); Primary Completion 2009-12-31 (Actual); Study Completion 2009-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (32):
- Belgium (32):
  - ASZ Aalst, Aalst
  - ZNA Middelheim, Antwerp
  - ZNA Stuivenberg, Antwerp
  - AZ Sint Lucas Brugge, Assebroek
  - CH EpiCURA Site Ath, Ath
  - CH EpiCURA Site Louis Caty, Baudour
  - Imeldaziekenhuis, Bonheiden
  - Clinique Saint-Jean- Botanique, Brussels
  - CHU Brugmann (Victor Horta), Brussels
  - Clin Univ de Bxl Hôpital Erasme, Brussels
  - HIS (Joseph Bracops), Brussels
  - UZ Brussel, Brussels
  - CHIREC Edith Cavell, Brussels
  - Cliniques Universitaires St-Luc, Brussels
  - CHU de Charleroi, Charleroi
  - AZ Sint Blasius (Dendermonde), Dendermonde
  - UZ Antwerpen, Edegem
  - ZOL (Sint Jan), Genk
  - AZ Sint Lucas (Sint Lucas), Ghent
  - UZ Gent, Ghent
  - CH EpiCURA Site Hornu, Hornu
  - CHR Hutois, Huy
  - Jan Yperman Onze Lieve Vrouw, Ieper
  - UZ Leuven Gasthuisberg, Leuven
  - Chr de La Citadelle, Liège
  - CHU Sart-Tilman, Liège
  - Clinique Saint-Joseph, Liège
  - AZ Delta (Campus Wilgenstraat), Roeselare
  - AZ Nikolaas (Sint Niklaas), Sint-Niklaas
  - CHWapi site IMC, Tournai
  - AZ Turnhout Sint Jozef, Turnhout
  - CHR de Verviers - East Belgium, Verviers

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Methoxy Polyethylene Glycol-Epoetin Beta
Started | 35
Completed | 21
Not Completed | 14
Not completed — Lost to Follow-up | 1
Not completed — Adverse Event | 2
Not completed — Death | 2
Not completed — Insufficient Therapeutic Response | 1
Not completed — Failure to Return | 1
Not completed — Dialysis Initiation | 5
Not completed — Blood Transfusion | 2

BASELINE CHARACTERISTICS:
Population: The safety population included all participants who received at least one dose of active drug.
Arm/Group | Methoxy Polyethylene Glycol-Epoetin Beta
Number analyzed (Participants) | 34
Age, Continuous [Median (Full Range); unit: years] | 77 [42 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 24

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Maintaining Average Hemoglobin Concentration During Efficacy Evaluation Period (EEP) Within Target Range
Description: The EEP was week 29 through week 36. The target range for average hemoglobin concentration was 10.0 - 12.0 g/dL.
Time Frame: Weeks 29-36
Population: Intent-to-Treat (ITT) population included all participants who entered the titration period and received active drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Methoxy Polyethylene Glycol-Epoetin Beta
Number analyzed (Participants) | 34
percentage of participants | 41 [24.7 to 59.3]

2. Secondary Outcome: Change From Baseline in Hemoglobin Concentration to Efficacy Evaluation Period (EEP)
Description: The mean change Baseline Hemoglobin to the time adjusted average of Hemoglobin during the EEP.
Time Frame: Weeks 0-36
Population: ITT population included all participants who entered the titration period and received active drug.
Measure: Mean (Standard Deviation); unit: grams/deciliter (g/dL)
Arm/Group | Methoxy Polyethylene Glycol-Epoetin Beta
Number analyzed (Participants) | 34
grams/deciliter (g/dL) | 0.99 (1.38)

3. Secondary Outcome: Percentage of Participants Maintaining Hemoglobin Concentrations Within Range of 10-12 Grams/Deciliter (g/dL) Throughout Efficacy Evaluation Period (EEP)
Time Frame: Weeks 29-36
Population: ITT population included all participants who entered the titration period and received active drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Methoxy Polyethylene Glycol-Epoetin Beta
Number analyzed (Participants) | 34
percentage of participants | 23.5 [10.8 to 41.2]

4. Secondary Outcome: Mean Time Spent in Hemoglobin Range of 10-12 g/dL During Efficacy Evaluation Period (EEP)
Time Frame: Weeks 29-36
Population: ITT population included all participants who entered the titration period and received active drug.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Methoxy Polyethylene Glycol-Epoetin Beta
Number analyzed (Participants) | 34
days | 28.6 (21.2)

5. Secondary Outcome: Percentage of Participants With Adverse Events
Description: An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.
Time Frame: Weeks 1-40
Population: The safety population included all participants who received at least one dose of active drug.
Measure: Number; unit: percentage of participants
Arm/Group | Methoxy Polyethylene Glycol-Epoetin Beta
Number analyzed (Participants) | 34
percentage of participants | 97

ADVERSE EVENTS:
Time Frame: Weeks 1-40
Arm/Group | Methoxy Polyethylene Glycol-Epoetin Beta
Serious Adverse Events (participants affected / at risk) | 15/34
Other Adverse Events (participants affected / at risk) | 29/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Methoxy Polyethylene Glycol-Epoetin Beta (N=34)
Anaemia (Blood and lymphatic system disorders) | 2
Pancytopenia (Blood and lymphatic system disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 2
Cardiac failure congestive (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Oesophagitis (Gastrointestinal disorders) | 1
Administration related reaction (General disorders) | 1
Asthenia (General disorders) | 1
Medical device complication (General disorders) | 1
Pyrexia (General disorders) | 1
Sudden cardiac death (General disorders) | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 1
Diarrhoea infectious (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Pseudomembranous colitis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Carotid artery stenosis (Nervous system disorders) | 1
Renal failure acute (Renal and urinary disorders) | 1
Renal failure chronic (Renal and urinary disorders) | 2
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1
Extremity necrosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Methoxy Polyethylene Glycol-Epoetin Beta (N=34)
Atrial fibrillation (Cardiac disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 2
Gastric ulcer (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 2
Oesophagitis (Gastrointestinal disorders) | 2
Chest pain (General disorders) | 2
Fatigue (General disorders) | 5
Oedema (General disorders) | 4
Bronchitis (Infections and infestations) | 6
Gastroenteritis (Infections and infestations) | 2
Nasopharyngitis (Infections and infestations) | 3
Fall (Injury, poisoning and procedural complications) | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2
Headache (Nervous system disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2
Hypertension (Vascular disorders) | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.